CLINICAL TRIAL: NCT07167758
Title: A Phase 2a, Randomized, Multicenter, Double-Blind, Placebo- Controlled Study to Evaluate the Efficacy, Safety, and Pharmacokinetics of Multiple Subcutaneous Doses of TRIV-509 in Adults With Moderate to Severe Atopic Dermatitis
Brief Title: A Study Evaluating TRIV-509 in Atopic Dermatitis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Triveni Bio (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 509-101
Record Dates: First submitted 2025-08-19; First posted 2025-09-11 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- First TRIV-509 then Placebo (Experimental)
  Interventions: Drug: TRIV-509; Drug: Placebo
- First Placebo then TRIV-509 (Experimental)
  Interventions: Drug: TRIV-509; Drug: Placebo

INTERVENTIONS:
Drug: TRIV-509 — TRIV-509 (Subcutaneous injection)
Drug: Placebo — Drug: Placebo (Matching Placebo subcutaneous injection)

SUMMARY:
The goal of this interventional study is to learn if TRIV-509 works to treat moderate to severe atopic dermatitis in adults. It will also evaluate the safety of TRIV-509.

Participants will receive 4 doses of the study intervention that they are randomized to (TRIV-509 or placebo), and at Week 16 will cross over and receive 4 doses of the other study intervention.

The study duration for individual participants is up to 57 weeks, including a Screening period of up to 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Has Atopic Dermatitis.
* Has moderate to severe, active and symptomatic AD

Exclusion Criteria:

* Severe or uncontrolled medical conditions.
* Use of topical treatments, phototherapy, systemic immunosuppressives or immunomodulatory therapies, or immunomodulatory biologics, within stated washout periods.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-08-26 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with improvement of AD at Week 16 | Baseline to Week 16

SECONDARY OUTCOMES:
Percentage of participants with improvement of AD at Week 16 | Baseline through Week 16
Percentage of participants with TEAEs. | For 16 Weeks
Percentage of participants with SAEs. | For 16 Weeks
Percentage of participants with anti-TRIV-509 antibodies | For 16 Weeks
Serum concentration of TRIV-509 | For 16 Weeks

CONTACTS AND LOCATIONS:
Locations (31):
- United States (14):
  - Triveni Bio Site #11, Fountain Valley, California
  - Triveni Bio Site #4, San Diego, California
  - Triveni Bio Site #3, Miami, Florida
  - Triveni Bio Site #7, Tampa, Florida
  - Triveni Bio Site #9, Tampa, Florida
  - Triveni Bio Site #6, Indianapolis, Indiana
  - Triveni Bio Site #10, South Bend, Indiana
  - Triveni Bio Site #1, Camp Hill, Pennsylvania
  - Triveni Bio Site #20, Pittsburgh, Pennsylvania
  - Triveni Bio Site #16, Bellaire, Texas
  - Triveni Bio Site #5, Dallas, Texas
  - Triveni Bio Site #2, Dallas, Texas
  - Triveni Bio Site #14, Springville, Utah
  - Triveni Bio Site #8, Spokane, Washington
- Canada (5):
  - Triveni Bio Site #13, Ajax, Ontario
  - Triveni Bio Site #17, Newmarket, Ontario
  - Triveni Bio Site #12, Niagara Falls, Ontario
  - Triveni Bio Site #15, North York, Ontario
  - Triveni Bio Site #19, Ottawa, Ontario
- Czechia (4):
  - Triveni Bio Site #22, Ostrava
  - Triveni Bio Site #31, Pardubice
  - Triveni Bio Site #21, Prague
  - Triveni Bio Site #23, Prague
- Poland (7):
  - Triveni Bio Site #28, Warsaw, Masovian Voivodeship
  - Triveni Bio Site #24, Chorzów, Silesian Voivodeship
  - Triveni Bio Site #25, Katowice, Silesian Voivodeship
  - Triveni Bio Site #27, Katowice, Silesian Voivodeship
  - Triveni Bio Site #30, Poznan, Wielkopolska
  - Triveni Bio Site #26, Poznan, Wielkopolska
  - Triveni Bio Site #29, Sosnowiec
- Triveni Bio Site #18, Kyiv, Ukraine

IPD SHARING:
Plan to Share IPD: No